CLINICAL TRIAL: NCT02518503
Title: Higher Potency Statins and the Risk of New Diabetes: Multicentre, Observational Study of Administrative Databases
Brief Title: High Potency Statins and the Risk of Diabetes
Acronym: Statins-DM
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q12-02
Record Dates: First submitted 2015-08-04; First posted 2015-08-07 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Disease
Keywords: Diabetes Mellitus; Statins; HMG-CoA reductase inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus | interventions — Rosuvastatin Calcium; Atorvastatin; Simvastatin; Fluvastatin; Pravastatin; Lovastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High potency statin users: Exposure will be defined as a new prescription for a high dose statin (high doses of rosuvastatin, high doses of atorvastatin, and high doses of simvastatin) between 1 January 1997 and 31 March 2011, or 1 year after the beginning of data availability.
  Interventions: Drug: Rosuvastatin (≥10 mg); Drug: Atorvastatin (≥20 mg); Drug: Simvastatin (≥40 mg)
- Low potency statin users: Exposure will be defined as a new prescription for a low dose statin (all doses of fluvastatin, all doses of pravastatin, all doses of lovastatin; low doses of atorvastatin and simvastatin) between 1 January 1997 and 31 of March 2011, or 1 year after the beginning of data availability.
  Interventions: Drug: Fluvastatin; Drug: Pravastatin; Drug: Lovastatin; Drug: Rosuvastatin (<10mg); Drug: Atorvastatin (<20mg); Drug: Simvastatin (<40 mg)

INTERVENTIONS:
Drug: Rosuvastatin (≥10 mg) — Current cumulative exposure to high dose rosuvastatin (ATC C10AA07) will be defined as a prescription for ≥10 mg of rosuvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-<365 days, or 366-730 days).
  Groups: High potency statin users
Drug: Atorvastatin (≥20 mg) — Current cumulative exposure to high dose atorvastatin (ATC C10AA05) will be defined as a prescription for ≥20 mg of atorvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-<365 days, or 366-730 days).
  Groups: High potency statin users
Drug: Simvastatin (≥40 mg) — Current cumulative exposure to high dose simvastatin (ATC C10AA01) will be defined as a prescription for ≥40 mg of simvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-<365 days, or 366-730 days).
  Groups: High potency statin users
Drug: Fluvastatin — Current cumulative exposure to fluvastatin (ATC C10AA04) will be defined as a prescription for any dose of fluvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-<365 days, or 366-730 days).
  Groups: Low potency statin users
Drug: Pravastatin — Current cumulative exposure to pravastatin (ATC C10AA03) will be defined as a prescription for any dose of pravastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-<365 days, or 366-730 days).
  Groups: Low potency statin users
Drug: Lovastatin — Current cumulative exposure to lovastatin (ATC C10AA02) will be defined as a prescription for any dose of lovastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-<365 days, or 366-730 days).
  Groups: Low potency statin users
Drug: Rosuvastatin (<10mg) — Current cumulative exposure to low dose rosuvastatin (ATC C10AA07) will be defined as a prescription for <10mg of rosuvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-<365 days, or 366-730 days).
  Groups: Low potency statin users
Drug: Atorvastatin (<20mg) — Current cumulative exposure to low dose atorvastatin (ATC C10AA05) will be defined as a prescription for <20 mg of atorvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-<365 days, or 366-730 days).
  Groups: Low potency statin users
Drug: Simvastatin (<40 mg) — Current cumulative exposure to low dose simvastatin (ATC C10AA01) will be defined as a prescription for <40 mg simvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-<365 days, or 366-730 days).
  Groups: Low potency statin users

SUMMARY:
Statins are a class of cholesterol lowering medications that are prescribed for the prevention and treatment of cardiovascular disease. The purpose of this study is to determine if there is an increased risk of new diabetes when exposed to high potency statins, compared to low potency statins, among patients who had a recent cardiovascular event or procedure.

The investigators will carry out separate population based cohort studies using administrative health care databases in eight jurisdictions in Canada, the US, and the UK. The cohort will be defined by the initiation of a statin, with follow-up until a diagnosis of incident diabetes or a prescription for insulin or an oral antidiabetic medication. The results from the separate sites will be combined in a meta-analysis to provide an overall assessment of the risk of new onset diabetes in subjects starting a statin.

DETAILED DESCRIPTION:
The study objective is to determine whether the use of high potency statins, compared with the use of low potency statins, is associated with an increased risk of incident diabetes following hospitalisation for a cardiovascular event or procedure. The investigators will use a common-protocol approach to conduct retrospective cohort studies using health care data from eight jurisdictions (the Canadian provinces of Alberta, Manitoba, Nova Scotia, Ontario, Quebec, and Saskatchewan, as well as the United States (US) MarketScan and the United Kingdom (UK) Clinical Practice Research Datalink [CPRD]). The Canadian provincial databases contain information on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs at a population level. The CPRD is a clinical database that is representative of the UK population and contains the records for patients seen at over 680 general practitioner practices in the UK; these data will be linked to the Hospital Episode Statistics (HES) database, which contains in-hospital diagnosis and procedure data. US MarketScan includes individuals and their dependents covered by large U.S. employer health insurance plans, and government and public organizations.

Study population

In each jurisdiction, the investigators will assemble a study cohort that includes all patients with a new prescription for a statin (after hospital discharge), including simvastatin, lovastatin, pravastatin, fluvastatin, atorvastatin, and rosuvastatin, from the earliest availability of data at each site to the last date of available data. The date of study cohort entry is defined by the prescription date of the newly-prescribed statin. Patients will be followed from the date of study cohort entry until an event (defined below) or censoring due to death, departure from the database, 24 months after the initiation of statin treatment, a dispensing for cerivastatin, or the end of the study period (31 March 2011 or the last date of data availability at that site), whichever occurs first. Data from Alberta, Ontario, and Nova Scotia will be restricted to patients aged 65 years and older as prescription data are not available for younger patients.

Case-control selection

The cohort defined above will be analyzed using a nested case-control analysis, where cases are defined as a hospitalization for incident diabetes or the prescription for an insulin or an oral antidiabetic medication. Risk set sampling will be used to randomly select up to 10 controls for each case, matched on sex, age (± two years; however, if no controls are available, within five years), and cohort entry (± 90 days).

Exposure assessment

The exposure categories will be separated by statin potency (high vs. low dose), and the duration of current exposure. For all cases and controls, exposure will be defined hierarchically; more specifically, patients who receive both a high and low potency statin within the same exposure category will be classified as high potency statin users. Current use of a high potency statin will be defined by the last prescription for a high dose statin prior to the index date. Current users will be further classified into three mutually exclusive durations of current exposure (≤120, 121-365, and 366-730 days).

Statistical analyses

Conditional logistic regression will be used to estimate the odds ratios and corresponding 95% confidence intervals (CIs) of the association between statin use and the diabetes endpoint, comparing current use of high potency statins to low potency statins. This is considered the primary analysis. Several sensitivity analyses will be performed to assess the robustness of study results and address some of the study limitations. High dimensional propensity scores will be estimated for all patients in the cohorts using logistic regression. Finally, all site-specific estimates will be meta-analyzed using fixed or random-effects models with inverse variance weighting. The amount of between-site heterogeneity will be estimated using the I square statistic.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital with a diagnosis (principal or secondary) for acute myocardial infarction or stroke or a procedure for coronary artery bypass graft or percutaneous coronary intervention during their stay in hospital, with no record of a diabetes diagnosis during their hospitalization
* Receipt of a prescription for a statin within 90 days of hospital discharge
* Patients who are at least 40 years of age at cohort entry
* Patients with at least one year of history in the database

Exclusion Criteria:

* Patients under the age of 40 (<66 in jurisdictions with drug data for seniors only)
* Patients with less than one year of history in the database
* Patients who received any cholesterol lowering drugs or diabetes medication/diagnosis in the previous year

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each jurisdiction, the investigators will assemble a study cohort that includes all patients with a new prescription for a statin, including simvastatin, lovastatin, pravastatin, fluvastatin, atorvastatin, and rosuvastatin between 1 January 1998 (or one year after the beginning of data availability) and 31 March 2011. The date of study cohort entry is defined by the prescription date of the newly-prescribed statin after hospital discharge.
Sampling Method: Probability Sample
Enrollment: 136966 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Incident type 2 diabetes | Patients will be followed from the date of study cohort entry until either hospitalization for diabetes or censoring (whichever occurs first), or will be assessed for up to 24 months.
  Patients with a first-hospitalization, receiving a principle or secondary diagnosis for diabetes (ICD-9: 250; ICD-10: E10, E11, E12, E13, E14), or a prescription for insulin or an oral antidiabetic medication.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Dormuth, M.Sc., Sc.D., Principal Investigator — Departments of Anesthesiology, Pharmacology and Therapeutics, University of British Columbia, Vancouver,BC

REFERENCES:
- [Result] Dormuth CR, Filion KB, Paterson JM, James MT, Teare GF, Raymond CB, Rahme E, Tamim H, Lipscombe L; Canadian Network for Observational Drug Effect Studies Investigators. Higher potency statins and the risk of new diabetes: multicentre, observational study of administrative databases. BMJ. 2014 May 29;348:g3244. doi: 10.1136/bmj.g3244. PMID 24874977
- See also: This organization's website describing general functions, other CNODES projects, and investigator profiles. — http://Info@cnodes.ca